CLINICAL TRIAL: NCT01026870
Title: A 12-Week Placebo-Controlled Efficacy and Safety Study of Mometasone Furoate Monotherapy in Subjects With Persistent Asthma Previously Treated With Low-Dose Inhaled Glucocorticosteroids
Brief Title: Efficacy and Safety of Mometasone Furoate for Persistent Asthma Previously Treated With Low-Dose Inhaled Glucocorticosteroids (ICS) (Study P06115)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06115
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate (MF) metered-dose inhaler 100 mcg BID (Active Comparator): 2 inhalations from a MF 50 mcg inhaler each morning and evening, approximately 12 hours apart, for 12 weeks
  Interventions: Drug: SCH 32088 mometasone furoate (MF) metered-dose inhaler
- Placebo metered-dose inhaler BID (Placebo Comparator): 2 inhalations from a matching placebo inhaler each morning and evening, approximately 12 hours apart, for 12 weeks.
  Interventions: Drug: Placebo metered-dose inhaler BID

INTERVENTIONS:
Drug: SCH 32088 mometasone furoate (MF) metered-dose inhaler — 2 inhalations from a MF 50 mcg inhaler each morning and evening, approximately 12 hours apart, for 12 weeks.
  Other Names: SCH 032088
  Arms: Mometasone furoate (MF) metered-dose inhaler 100 mcg BID
Drug: Placebo metered-dose inhaler BID — 2 inhalations from a placebo metered-dose inhaler each morning and evening, approximately 12 hours apart, for 12 weeks.
  Arms: Placebo metered-dose inhaler BID

SUMMARY:
Mometasone furoate (MF) is a synthetic glucocorticosteroid that, when administered to asthma patients with a dry powder inhaler (Asmanex® Twisthaler®) at dosages of 100 to 400 mcg twice daily, has been shown to improve lung function, reduce symptoms of asthma, and reduce frequency and severity of exacerbations by reducing airway inflammation, with a relatively low potential to cause systemic side effects such as hypothalamic-pituitary-adrenal (HPA) axis suppression.

An experimental formulation of MF 100 mcg delivered twice daily via a pressurized metered-dose inhaler (MDI) also has been shown to be effective in improving lung function of asthma patients as measured by forced expiratory volume in 1 second (FEV1). This trial is designed to verify the effectiveness of twice daily MF MDI 100 mcg in treating asthma in adults and adolescents previously treated with low dosages of inhaled corticosteroids (ICS), as measured by improvement in morning FEV1 and time to first asthma exacerbation over 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* An adult or adolescent subject with a diagnosis of persistent asthma of >=6 months duration may be selected for this study.
* Both subject (and/or parent/guardian, if appropriate) and investigator must agree that changing therapy is acceptable and poses no inherent risk.
* Subject must have been using a low daily maintenance dose of inhaled corticosteroids (ICS), with or without added long-acting β2-agonist (LABA), for >=12 weeks prior to Screening, and must have been on a stable regimen (daily dose unchanged) for at least the last 2 weeks of that period.
* At Screening, the subject must have a prebronchodilator FEV1 between 60% and 90% of the predicted value when restricted medications have been withheld.
* To be randomized, the subjects must be symptomatic with FEV1 at Baseline must be between 50% and 85% of predicted.

Exclusion Criteria:

* A subject must not have been admitted to the hospital for management of airway obstruction within the last 3 months prior to Screening, and must not have experienced an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication, as judged by the clinical investigator at any time from Screening to Baseline/Randomization.
* In addition, a subject must not have demonstrated a decrease in absolute FEV1 of >20% at any time from Screening to Baseline, or a decrease in AM peak expiratory flow (PEF) below the PEF stability limit on any 2 consecutive days prior to Baseline/Randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Endpoint in the morning (AM trough) forced expiratory volume in 1 second (FEV1) | Endpoint: last non-missing post-Baseline observation carried forward over 12 weeks of treatment

SECONDARY OUTCOMES:
Time to first severe asthma exacerbation during the 12 week Treatment Period | 12 weeks